CLINICAL TRIAL: NCT00578435
Title: Allogeneic Bone Marrow Transplantation for the Treatment of Genetic Disorders of Erythropoiesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Fourid Boulad, Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-005
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Genetic Disorders; Sickle Cell Anemia
Keywords: ERYTHROPOIESIS; Genetic Disorders; Sickle Cell Anemia; Thalassemia; Diamond Blackfan Anemia
MeSH Terms: conditions — Genetic Diseases, Inborn; Anemia, Sickle Cell; Thalassemia; Anemia, Diamond-Blackfan | interventions — Busulfan; Cyclophosphamide

INTERVENTIONS:
Procedure: Busulfan, Cyclophosphamide, BMD — Busulfan 0.8 or 1 mg/Kg/day Days 8-6 Cyclophosphamide 50 mg/Kg/day Days 2-5 BMT Day 0

SUMMARY:
The purpose of this study is to determine and confirm the role of bone marrow transplantation in the treatment of disorders of the red cell and hemoglobin including sickle cell anemia, thalassemia and diamond blackfan anemia.

DETAILED DESCRIPTION:
The trial proposed is a single armed phase II treatment protocol designed to examine the engraftment,toxicity and graft-versus-host disease following a novel cytoreductive regimen including cyclophosphamide and Busulfan for the treatment of patients with Severe Sickle Cell Anemia,Thalassemia, and Diamond Blackfan Anemia using stem cell transplants derived from HLA-genotypically identical siblings.

Patients will be conditioned for transplantation with cyclophosphamide (50 mg/kg/day x 4 days), and busulfan [(if < 4 years of age 1 mg/kg 4 times per day x 4 days), (if > 4 years of age 0.8 mg/kg 4 times per day x 4 days)]. Patients will receive Methotrexate & Cyclosporin-A for prophylaxis against GvHD and GCSF to promote engraftment.

The preferred source of stem cells from related HLA-matched related donors will be unmodified bone marrow stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe HOMOZYGOUS SICKLE CELL ANEMIA or SICKLE/BETA THALASSEMIA
* Neurologic event (stroke or hemorrhage).
* Abnormal cerebral MRI scan and cerebral arteriogram or MRI angiographic study (MRA) and impaired neuropsychologic testing.
* Recurrent acute chest syndrome (> 2 episodes)
* Stage I-II sickle chronic lung disease
* Sickle cell nephropathy (moderate or severe proteinuria or GFR 30-50% of predicted for age.
* Major visual impairment in at least one eye with bilateral proliferative retinopathy.
* Osteonecrosis of multiple bones
* Chronic debilitating pain secondary to vasoocclusive crisis (>= 3 episodes per year for >= 3 years) Recurrent priapism
* Allo-immunization with the development of antibodies following chronic transfusion therapy
* Patients with HOMOZYGOUS SICKLE CELL ANEMIA or SICKLE/BETA THALASSEMIA with the following criteria will be considered for accrual on this protocol
* Patients < 2 years with high WBC counts and/or >1 episode of dactylitis and/or a Hgb < 7 g/dl
* History of death from sickle cell disease in sibship of patient
* Patients with BETA-THALASSEMIA MAJOR with Lucarelli class 1 or 2 risk status i.e with only 0-2 of the following factors: hepatomegaly, portal fibrosis, or poor chelation therapy
* Patients with DIAMOND-BLACKFAN ANEMIA who have failed conventional therapy.
* Patients must have an HLA-compatible related donor. The donor must be healthy and able to undergo general anesthesia. Donors with heterozygous sickle cell anemia (hemoglobin AS) or with heterozygous thalassemia are acceptable donors.
* At the time of referral for transplantation, patients must be in good clinical condition without any evidence of infections and a Karnofsky or Lansky pediatric performance scale > 70%
* Each patient and donor must be willing to participate as a research subject and must sign an informed consent form after having been advised as to the nature and risk of the study prior to entering the protocol. Parents or legal guardians of patients who are minor will sign the consent form after being advised of the nature and risks of the study

Exclusion Criteria:

* Patients whose life expectancy is less than 8 weeks. Patients with a Karnofsky or Lansky performance score of < 70%
* Patients with severe major organ dysfunction:
* Patients with severe renal impairment. This will be determined by a creatinine clearance < 70 ml/min/1.73 m2 (or serum creatinine > 1.5 x Normal) or by a glomerular filtration rate < 30% of predicted normal for age
* Inadequate cardiac function as determined by fractional shortening < 28% on echocardiogram, and/or ejection fraction of < 50% on echocardiogram or RNCA.
* Patients with FS of 23-28% who show an increase in FS in response to stress on the supine bicycle ergometer are eligible
* Major liver dysfunction: SGOT > 3 x upper limit of normal. Hyperbilirubinemia will not be used as an exclusion criteria because of the hemolytic component of the bilirubin. Patients with active hepatitis or severe liver fibrosis will also be excluded
* Severe residual functional neurologic impairment
* Stage III-IV sickle chronic lung disease
* Pregnant or lactating women are excluded

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1994-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Define the role of bone marrow transplantation for the treatment of sickle cell disease and the reversibility of sickle cell vasculopathy and organ damage, good risk thalassemia major and Diamond-Blackfan Anemia. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Farid Boulad, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org